CLINICAL TRIAL: NCT05513534
Title: The Effects of Yoga and Power Training on Mindfulness, Psychological Wellbeing, and Functional Ability of Individuals With Parkinson's Disease.
Brief Title: Mindfulness and Yoga or Resistance Exercise Training Fpr Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220477
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Resistance Training; Yoga
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: We will compare Yoga and circuit resistance tarining impacts on mindfulness, anxiety, cognition, muscle structure, and physical performance in people with Parkinson's disease.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be masked concerning the intervention provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Hatha Yoga (Experimental): A yoga program adapted for those with PD will be used in the current study. It will be conducted over a 16-week period and consists of twice-weekly sessions lasting approximately one hour. The program will be based on principles of Hatha yoga which incorporate longer holds and deep breathing. Each session will include a warm-up, three yoga flows, a balance training section, and a cooldown phase. The first four weeks will emphasize proper alignment, breathing, and technique. Additionally, the classes will be led by a certified yoga instructor and include multiple on-site assistants to ensure a safe training environment. Participants will also be provided with assistive devices (i.e. chairs, yoga blocks, and blankets) if they are required.
  Interventions: Other: Yoga
- Power Resisatnce Training (Experimental): : A high-velocity resistance (power) will be conducted over a 16-week period and consists of twice-weekly sessions lasting approximately one hour. Each training session will begin with a brief warm-up. Each session will consist of three sets of 10 repetitions each with 1.5 to 2- to minute rest periods between sets. Participants will be instructed to control the concentric and eccentric velocity of each exercise, with each phase lasting approximately two to three seconds. Exercise order will be randomized during each session and upper and lower body exercises will be alternated whenever possible.
  Interventions: Other: High-speed Resistance Training

INTERVENTIONS:
Other: Yoga — A standard yoga program will be provided using Hatha poses.
  Arms: Standard Hatha Yoga
Other: High-speed Resistance Training — Each session will consist of three sets of 10 repetitions each with 1.5 to 2-minute rest periods between sets. Participants will be instructed to control the concentric and eccentric velocity of each exercise, with each phase lasting approximately two to three seconds
  Arms: Power Resisatnce Training

SUMMARY:
The investigators propose to compare the effects of a 16-week specially designed yoga program to a power-based resistance training program on affect trait mindfulness, anxiety, depression, functionality, and quality of life. As secondary measures, we propose to compare the effects of these exercise programs on measures of executive function (EF), sleep, disease stage, motor symptoms, muscle quality, rigidity, strength, power, and mobility.

DETAILED DESCRIPTION:
Yoga has long been recognized as a therapeutic intervention for improving mindfulness and psychological well-being. Yoga represents a unique exercise activity that employs mindfulness-based practices and various balance postures to improve physical and mental health. Yoga is a gentle form of exercise that can be easily adapted to populations suffering from physical and mental limitations and has been shown to improve physical and psychological functioning in individuals with PD. Though research continues to support the positive psychological effects of yoga, it is unclear whether this is due to the unique mindfulness-rooted approach of yoga or general increases in physical activity.

Power-based resistance training has had promising results in the PD community. Improvements in balance, gait, and increases in leg muscle power and strength have been shown in PD patients after power training interventions. Although power training is a beneficial exercise modality in the treatment of motor symptoms, the effects of power training on nonmotor symptoms have yet to be established.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with mild to moderate PD [Hoehn and Yahr (H&Y) stage 1-3];
* over 50 years of age;
* stable use of medication;
* able to walk 15 m independently with or without an assistive device;
* the ability to get up and down from the floor with minimal assistance;
* not currently participating in yoga or resistance training more than one time per week;
* able to understand and communicate in English; and,
* able to provide informed consent.

Exclusion Criteria:

* cognitive impairment as designated by a score of less than 23 on the Montreal Cognitive Assessment (MoCA)]; and,
* any clinically significant medical condition, such as cardiopulmonary disease and musculoskeletal problems. Subjects providing affirmative answers on a Physical Activity Readiness Questionnaire (PAR-Q) or Health Status Questionnaire related to cardiopulmonary disease or musculoskeletal impairments will be required to present a physical activity clearance from their physician.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire (PDQ-39) | 15 minutes
  The PDQ-39 is one of the most widely used self-reported questionnaires designed to assess QoL in Parkinson's patients. It is composed of 39 items which are distributed over 8 separate scales including mobility, activities of daily living, emotional wellbeing, stigma, social support, cognition, communication, and bodily discomfort (Jenkinson et al., 1997). All items are answered on a 5-point Likert type scale (0= never, 1=occasionally, 2=sometimes, 3=often, 4=always). In addition, a summary index can be computed to assess the overall impact of PD on the responder.
Parkinson Anxiety Scale (PAS) | 2 minutes
  The Parkinson Anxiety Scale (PAS) is a frequently used observer or patient-rated anxiety measurement tool designed specifically for PD patients. The exam consists of three sub-scales for persistent anxiety (dimension A), episodic anxiety (dimension B), and avoidance behavior (dimension C), with 5, 4, and 3 items, respectively. All items are scored on a 5-point Likert type scale (0=not or never, 4=severe or almost always). A cut-off point of 14 is optimal to detect anxiety. Self-administered, the test takes approximately 2 minutes.
Beck Depression Inventory | 5 minutes
  The Beck Depression Inventory is a widely used self-report inventory to assess the severity of depressive symptoms in adults in the past two weeks. The BDI-II has been validated in patients with PD. It includes both cognitive and somatic symptoms of depression and consists of 21 items using a 4-point Likert scale. A maximum score is 63 with 0-13 indicating none or minimal range depression, 14-19 mild, 20-28 moderate, and 29-63 severe.
Mindful Attention Awareness Scale (MAAS) | 5 minutes
  The Mindful Attention Awareness Scale is a single-factor measure of trait mindfulness comprised of 15 items. The scale evaluates attentiveness and awareness of the present moment with higher scores indicating a greater degree of mindfulness trait. All questions are answered on a 6-point Likert scale with a range from 1 to 6. The total possible score is 90 points with a minimum score of 15

SECONDARY OUTCOMES:
One-repetition maximum (1RM) testing | 10 minutes
  One-repetition maximum (1RM) strength testing will include leg press and chest press. After a warm-up, the subject do 10 repetitions a low resistance. The test will begin using a weight near the predicted maximum. The weight will then be increased or decreased depending on the subject's ability to perform the repetition using correct technique.
Timed Up & Go (TUG) | 3 minutes
  The TUG is a widely used clinical assessment for measuring fall risk and functional mobility. The test begins with participants sitting with their spines against a chair back and their hands on their laps. Upon verbal cue, subjects stand up, walk around a cone placed three meters from the front edge of the chair and then return to their seated position. The participants will be timed as they complete the task as quickly as possible. Each participant will perform one familiarization trial and two test trials, with at least a one-minute recovery between trials.
Quantitative Gait Assessment | 5 minutes
  Three-dimensional movement analysis of subjects gait patterns during a 10-meter walk.
Isokinetic Testing | 30 minutes
  The Biodex 4 Dynamometer will be used for all isokinetic testing. Subjects will be asked to perform an isokinetic warm-up of 10 repetitions of leg extension at 270 deg/s, be given a three-minute recovery, and then perform three maximal isokinetic quadriceps extensions at 90, 180, and 300 degrees/second using 2-minute recoveries in between sets. All results will be recorded. The repetitions producing the highest peak torque among the three efforts, and the average power for the repetitions will be used for statistical evaluation. Given the nature of isokinetic testing the resistance is at the speeds we have chosen, far below maximum.
Ultrasound | 20 minutes
  Ultrasound images of the quadriceps femoris muscle (vastus medialis, vastus lateralis, vastus intermedius, rectus femoris) will be taken on the thigh at the two-thirds and midpoint of the length between the anterior superior iliac spine and the upper border of the patella. A LOGIQ P9 R3 Ultrasound System (GE Healthcare, Buckinghamshire, UK) and 3-12 MHz linear array transducer probe will be used, and testing will be conducted on a padded treatment table. Care will be taken to maintain the same standardized body positions and probe locations for all participants. Minimal pressure will be applied by the researcher to reduce any tissue compression that would artificially influence the results. Before acquiring measurements, subjects will rest on the examination table for five minutes to avoid any potential movement-induced stiffness. To improve acoustic contact between the probe and skin, a water-soluble transmission gel will be used on the head of the probe.
Power Testing | 15 minutes
  ower testing will begin with a warm-up of 10 repetitions at 30% 1RM, followed by a 1-minute recovery period. A second warm-up of 5 repetitions at 30% 1RM will then be performed as rapidly as possible. Peak muscle power will then be assessed at 8 relative intensities (40, 50, 60, 70, and 80% 1RM) on the same resistance machines used for strength testing. The percentages will be randomized to reduce any order effect. For each repetition, the concentric phase will be performed as fast as possible, and the eccentric phase will be performed over 2-3 seconds. Each repetition will be verbally cued "3.2.1. Go!" This testing protocol is commonly used for power testing.34,35 Any repetition not performed properly will be repeated after a 1-minute break. Power output will be recorded from the display of each machine and cross-referenced with the electronic spreadsheets.
The Stroop Color Word Test | 5 minutes
  The Stroop color word test is another commonly used neurophysiological assessment which evaluates the participant's ability to inhibit cognitive inference. This cognitive domain is associated with EF and involves the processing of a stimulus where one feature of a previous stimulus may affect the simultaneous processing of a new stimulus. Typically, the test requires an individual to name the color of ink of color words printed in incongruent colors (incongruent condition), for example, the word "red" is printed in green ink. Participants must also complete a control task, where they read a color name printed in black ink and identify colored rectangles that correspond to that color as quickly as possible (congruent condition).
Trail-making Test (TNT) | 5 minutes
  The TMT is yet another frequently used neurophysiological assessment which examines visuospatial abilities, working memory and task switching abilities associated with executive function domains. The test is separated into two different assessments, part A and part B. Both tasks incorporate 25 circles distributed across a white sheet of paper. In part A, the circles are numbered from 1 to 25. In part B, the participant is presented with alternating numbers and letters. Both tasks require the participant to connect the circles with lines in ascending order as quickly as possible. It has been shown that TMT Part A is associated with EF domains of visuospatial abilities, whereas part B is associated with working memory and response inhibition. Those with PD have demonstrated decreased scores on both the TMT part A and B indicating executive function decrements.
Home Sleep Testing | 8 hours
  Study participants will have a home sleep study using the NoxA1 system that allows for monitoring of sleep (i.e., EEG) along with respiratory effort and oxygen saturation. The goal of the home sleep study is to exclude other respiratory-related sleep disorders.
Actigraphy | 168 hours
  An actigraph will be worn on the wrist for seven consecutive 24-hour periods, to collect data on habitual sleep duration. Wrist actigraphy is a technique for measuring movement over an extended recording period (days to weeks). Data garnered from wrist actigraphy will be used to derive variables such as habitual total sleep time, number and duration of awakenings per night, and napping behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No